CLINICAL TRIAL: NCT03804489
Title: Using "Decision Aids" to Help the Infant Family to Decide Whether the Baby Will Receive the Self-paid Oral Rotavirus Vaccine: A Randomized Controlled Trial.
Brief Title: Using "Decision Aids" to Help the Infant Family to Decide the Use of Oral Rotavirus Vaccine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Chieh Lin, Medical attending doctor, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 108HHC-03
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Rotavirus Vaccines
Keywords: Decision Aids; Shared decision making; Rotavirus Vaccines
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Decision aids
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision aids group (Experimental): Shared decision making using decision aids,
  Interventions: Other: Decision aids
- Control group (No Intervention): Standard oral explanation with booklet.

INTERVENTIONS:
Other: Decision aids — Decision aids in helping the infant family to decide whether the infant will or will not receive the oral rotavirus vaccine.
  Arms: Decision aids group

SUMMARY:
Using decision aids (DA) is one way to provide information to infant family and to involve them in making decisions about their baby's vaccination. We developed a DA administered after consultation for baby's family deciding on whether the baby will receive the self-paid oral rotavirus vaccine

DETAILED DESCRIPTION:
Background:

Acute gastroenteritis is one of the most common infectious diseases and still a major cause of pediatric morbidity and mortality worldwide. Rotavirus was still the major cause of acute gastroenteritis in infants and young children worldwide, including in Taiwan. The World Health Organization has recommended rotavirus vaccine, which became available in 2006, for all countries. However, not all of children in Taiwan received rotavirus vaccination. Using decision aids (DA) is one way to provide information to infant family and to involve them in making decisions about their baby's vaccination. We developed a DA administered after consultation for baby's family deciding on whether the baby will receive the self-paid oral rotavirus vaccine Patients and Methods Decision aids are interventions designed to help infant family make choices among options by providing information relevant to oral rotavirus vaccine. Infant coming to receiving regular routine vaccination at 1 month old are randomly assigned to receive a DA or the standard oral conversation (control condition) after the initial consultation. Infant family complete interview-based questionnaires 1 month later when they came back to hospital receiving 2-month-old regular routine vaccination and decide to receive self-paid oral rotavirus vaccine or not at that time. Primary outcome measures: decisional conflict and decision-making difficulties at 2-month-old.

Results and Conclusion The DA group are predicted to lower decisional conflict scores when compared with the control group. Our study hopes to support the efficacy of DA in helping the infant family to decide whether the baby will receive the self-paid oral rotavirus vaccine.

ELIGIBILITY:
Inclusion Criteria:

The one-month-old baby's family whose age is between 20 and 80 years old.

Exclusion Criteria:

1. . The doctor determines that the baby's family is not suitable; if baby's family cannot understand Chinese languages what we said.
2. . The participants' baby who have fever or contraindication for oral rotavirus.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-01-25 (Estimated); Primary Completion 2019-10-25 (Estimated); Study Completion 2019-12-25 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict | An average of 1 month after intervention
  Total score of decisional conflict scale
Decision-making difficulties | An average of 1 month after intervention
  Total score of decision-making scale

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Chieh Lin, MD, Principal Investigator — Department of Pediatrics, Shuang Ho Hospital, Taipei Medical University
Locations (1):
- Sheng-Chieh Lin, New Taipei City, No.291, Zhongzheng Road, Zhonghe District, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lin SC, Tam KW, Yen JY, Lu MC, Chen EY, Kuo YT, Lin WC, Chen SH, Loh EW, Chen SY. The impact of shared decision making with patient decision aids on the rotavirus vaccination rate in children: A randomized controlled trial. Prev Med. 2020 Dec;141:106244. doi: 10.1016/j.ypmed.2020.106244. Epub 2020 Sep 4. PMID 32891678